CLINICAL TRIAL: NCT07394803
Title: Physical Activity and Pregnant Women at Increased Social Risk: a Feasibility Study
Acronym: ACTIVA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Universidad Politecnica de Madrid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR(AMI)508/2024
Record Dates: First submitted 2026-01-14; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy
Keywords: physical activity during pregnancy; social risk; mental health; moderate physical activity; Facilities and barriers for physical activity in pregnant women
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Non-randomized multicenter feasibility trial will be performed piloting several components of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant individuals participating in the moderate physical activity program (Experimental): The design of the physical exercise program is supported by the Canadian and Spanish Guidelines (5,6,14) , for exercise throughout pregnancy and published by Barakat model (15) , supporting a minimum of 150 minutes per week of moderate intensity exercise. The program consists of three weekly sessions. The duration of every session lasts 55-60 minutes.
  Once a week, the Borg Scale of Perceived Effort is administered to participants, in order to have a more reliable assessment of the intensity of the activities, 12-14 (moderate; out of a 20-point scale) is the level used. The minimum adherence required for the participants will be 70% of the total sessions, but no restriction will be taken to the classes. The adherence to the program will be recorded.
  The intervention program will follow Barakat´s Model and consist three weekly sessions of 60 minutes, following a hybrid program (on-site and online via Zoom®). The on-site sessions will be held at CAP San Andreu in a gym room.
  Interventions: Behavioral: Moderate physical activity

INTERVENTIONS:
Behavioral: Moderate physical activity — The intervention program will follow a physical exercise program supported by the Canadian and Spanish Guidelines, for exercise throughout pregnancy and published by Barakat model, supporting a minimum of 150 minutes per week of moderate intensity exercise. It consists on three weekly sessions of 60 min, following a hybrid program (on-site and online via Zoom®). The on-site sessions will be held at CAP San Andreu in a gym room.
  Once a week, the Borg Scale of Perceived Effort is administered to have a more reliable assessment of the intensity of the activities, 12-14 (moderate; out of a 20-point scale) is the level used. The minimum adherence required for the participants will be 70% of the total sessions, but no restriction will be taken to the classes, adherence will be recorded.
  Women accepting participation, with no contraindications to perform physical activity, will sign the consent form- Implementation of the PA Program crossingbox that includes the physical activity program.

SUMMARY:
Objective: To test the feasibility of the implementation of a moderate intensity physical activity program during pregnancy in a group of pregnant women at social risk.

Methods: a non-randomized feasibility study piloting several components of the trial Inclusion criteria: > 18 yo, antenatal care at HVH and/or ASSIR SAP Muntanya, and vulnerable socioeconomical conditions.

Exclusion criteria: contraindications for the practice of physical activity during pregnancy according to Spanish and Canadian Guidelines.

Practical Course of the research: Women will be recruited for the study and will perform a physical activity moderate intensity hybrid (on-site and online) program during pregnancy (3 times per week 60 min sessions) and will respond to several questionnaires (Barriers, IPAQ, WHO-5, EPDS, STAI, SF-12, MOSSS, PSQI) Those who reject to participate in the program, will be offered to respond to these questionnaires. Main outcomes are the acceptability to the program, the reasons for rejection, the physical activity level during pregnancy, the barriers and facilitators to physical activity during pregnancy.

Number of recruiting centers: Hospital Vall d´Hebron and Primary Care Center ASSIR Muntanya (Centro de atención a la salud sexual y Reproductiva) Barcelona Nord.

Sample size: 60 aiming to achieve 30 women in the physical activity program

Statistical analyses: quantitative descriptive analysis.

Source of funding: no funding available, pending for funding

DETAILED DESCRIPTION:
Main objective: To test the feasibility of the implementation of a moderate intensity physical activity program during pregnancy in a group of pregnant women at social risk.

Specific objectives:

* To evaluate the acceptability of the physical activity program
* To evaluate barriers, facilitators and attitudes towards physical activity in relationship to the physical activity in this target group of population.
* To evaluate the level of physical activity achieved by this group of population during pregnancy, as well as the sedentarism.
* To evaluate the impact on the well-being and mental health of a moderate intensity physical activity program during pregnancy in this target group of population.
* To evaluate the impact on physical health and perception of quality of life and sleep of a moderate intensity physical activity program during pregnancy in this target group of population.

Methods: a non-randomized feasibility study piloting several components of the trialI.

The inclusion criteria are: > 18 yo, antenatal care at HVH and/or ASSIR SAP Muntanya, and vulnerable socioeconomical conditions, according to the local antenatal protocol.

The exclusion criteria are the presence of contraindications for the practice of physical activity during pregnancy according to Spanish and Canadian Guidelines.

Practical Course of the research: Women will be recruited for the study and will perform a physical activity moderate intensity hybrid (on-site and online) program during pregnancy (3 times per week 60 min sessions), following the Barakat Model.

Pregnant individuals who are not interested and reject to participate will be offered to complete several questionnaires during pregnancy to better understand how active they are during pregnancy and what are the reasons to understand why they are not active, as well as the barriers and facilitators, and the perceptions of physical activity during pregnancy.

Main outcomes are the acceptability to the program, the reasons for rejection, the physical activity level during pregnancy, the barriers and facilitators to physical activity during pregnancy.

Secondary outcomes include:

* Mental Health outcomes: Wellbeing, Depression, Anxiety, Perceived stress, Health related quality of life (HRQoL), Sleep quality , Social support
* Physical health outcomes: Lumbar and pelvic pain through the pregnancy, Maternal weight gain during pregnancy and Pregnancy complications (preterm birth, gestational diabetes, pregnancy induced hypertension, low birth weight )

Questionnaires:

Barriers ( self-created), IPAQ, WHO-5, EPDS, STAI, SF-12, MOSSS, PSQI, PSS

Number of recruiting centers: Hospital Vall d´Hebron and Primary Care Center ASSIR Muntanya (Centro de atención a la salud sexual y Reproductiva) Barcelona Nord.

Sample size: 60 aiming to achieve 30 women in the physical activity programStatistical analyses: quantitative descriptive analysis.

Source of funding: no funding available, pending for funding

ELIGIBILITY:
Inclusion Criteria:

* Maternal age above 18 years old.
* Antenatal care at ASSIR Barcelona Nord (SAP Muntanya), and/or Hospital Vall d´Hebron.
* Fulfilling social risk criteria defined by the Local Protocol (13), that includes as vulnerable socioeconomical conditions: low economic income, unemployed, poor nutrition, low educational level, difficult access to perinatal healthcare and lack of social and familiar support.

Exclusion Criteria:

* Contraindications for the practice of physical activity during pregnancy according to the Spanish and/or Canadian (5,6,14)guidelines of physical activity during pregnancy (ref).
* Unable to communicate in the official language (Spanish or Catalan)
* Aiming to give birth in a different setting of the study setting.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability | "Baseline"
  Number of individuals that agrees to participate in the study at "baseline", after offering the study participations and explaining the study procedure, and sign the informed consent document
Rejection to participate in the physical activity program | "Baseline"
  Number of individuals that reject to participate in the study at "baseline" after explaining the study procedure and signed rejection CI
Reasons for rejection | "Baseline"
  - Reason for rejection to participate in the study: lack of time, cultural, stigma related mental health or physical activity, hesitance regarding participation on a trial, others... when offering the study participation at baseline
Perceived barriers for performing physical activity during pregnancy | "through study completion, an average of 1 year"
  A Likert Scale questionnaire self-created will be assessed by each participant (23 items will be assessed)
Adherence to the program | "through study completion, an average of 1 year"
  Registration of the attendance to the on-site PA classes will be mandatory, and also in the online (via Zoom), it will be assesed.

SECONDARY OUTCOMES:
Well-being | At enrollment, end of pregnancy and 4-6 weeks postpartum
  Using the WHO-5 questionnaire. Raw scores ranging from 0 (minimum, worst imaginable well-being) to 25 (maximum, best imaginable well-being)
Lumbar and pelvic pain | 1 year
  Lumbar and pelvic pain through the pregnancy will be assessed during pregnancy medical records yes/no
maternal weight gain during pregnancy | from enrollment to 1 month postpartum
  Maternal weight gain in Kg during antenatal care
Depression symptoms | At enrollment, end of pregnancy and at 4-6 weeks postpartum
  EPDS questionnaire, ranges from a total score of 0 and a maximum total score of 30. Each item is scored from 0 to 3, with higher scores indicating more severe depressive symptoms
Anxiety symptoms | At enrollment, end of pregnancy and at 4-6 weeks postpartum
  STAI questionnaire ( trait-state). Consists of two 20-item subscales (State and Trait), each with a minimum score of 20 and a maximum score of 80. Higher scores indicate greater anxiety levels
Stress | At enrollment, end of pregnancy and at 4-6 weeks postpartum
  PSS questionnaire. The Perceived Stress Scale (PSS-10) ranges from 0 to 40, with 0 being the minimum (no stress) and 40 being the maximum (very high stress)
Health Related Quality of Life | At enrollment, end of pregnancy and at 4-6 weeks postpartum
  SF 12 questionnaire. The SF-12 health survey uses norm-based scoring, resulting in Physical (PCS) and Mental (MCS) Component Summary scores with a mean of 50 and a standard deviation of 10 in the general population. Scores generally range from approximately 0 to 100, where higher values indicate better health
Quality of Sleep | At enrollment, end of pregnancy and at 4-6 weeks postpartum
  Pittsburgh Sleep Questionnaire ( PSQI). The Pittsburgh Sleep Quality Index (PSQI) total global score ranges from a minimum of 0 to a maximum of 21. A lower score (0-5) indicates better sleep quality, while a higher score (>5) indicates poorer sleep quality
Social Support | At enrollment, end of pregnancy and at 4-6 weeks postpartum
  MOSSS questionnaire. The MOS Social Support Survey (MOS-SSS) typically uses 19 items rated on a 5-point Likert scale (1=None of the time to 5=All of the time), resulting in a minimum raw score of 19 and a maximum of 95. These scores are commonly transformed to a 0-100 scale, where 0 represents the lowest and 100 the highest possible social support
Physical Activity | At enrollment, end of pregnancy and at 4-6 weeks postpartum
  IPAQ questionnaire. The International Physical Activity Questionnaire (IPAQ) measures activity in MET-minutes/week, with categorizations for low (<600), moderate (600-3000), and high (>3000) levels. Data is cleaned by truncating daily activity to 180 minutes and requires activities to last at least 10 minutes. The minimum is 0, while high-level, vigorous activity can exceed 3000+ MET-min/week
Pregnancy complications: preterm birth | birth
  Gestational age at birth below 37 w
Pregnancy Complications: Gestational diabetes | during pregnancy, , both between 24-28 weeks
  Gestational diabetes, as 100 mg Glucose Tolerance Test positive or HbA1c> 5.7%
Birth Outcomes: Birth weight | 1 month
  Birth weight in Kg
Birth Outcomes: NICU admission | 1 month
  NICU Admission yes/no
Birth Outcomes | 1 month
  Apgar Score at birth 1/5/10 minutes
Pregnancy Complications: Pregnancy Induced Hypertension | during pregnancy and at birth
  Preeclampsia, Gestational Hypertension, Eclampsia and/or Placental Insuficiency ( IUGR)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Barakat, PhD, Study Director — Universidad Politécnica de Madrid, Spain
Locations (2):
- Spain (2):
  - Centros de Atenció a la salut sexual i reproductiva (ASSIR) in Barcelona Nord, Barcelona
  - Hospital Vall d´Hebron, Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided
Data could be shared upon request, and if ethical committe approves the sharing, and participants consent for the data sharing

REFERENCES:
- [Background] Wang E, Glazer KB, Howell EA, Janevic TM. Social Determinants of Pregnancy-Related Mortality and Morbidity in the United States: A Systematic Review. Obstet Gynecol. 2020 Apr;135(4):896-915. doi: 10.1097/AOG.0000000000003762. PMID 32168209
- [Background] Mottola MF, Davenport MH, Ruchat SM, Davies GA, Poitras VJ, Gray CE, Jaramillo Garcia A, Barrowman N, Adamo KB, Duggan M, Barakat R, Chilibeck P, Fleming K, Forte M, Korolnek J, Nagpal T, Slater LG, Stirling D, Zehr L. 2019 Canadian guideline for physical activity throughout pregnancy. Br J Sports Med. 2018 Nov;52(21):1339-1346. doi: 10.1136/bjsports-2018-100056. PMID 30337460
- [Background] Davenport MH, Ruchat SM, Poitras VJ, Jaramillo Garcia A, Gray CE, Barrowman N, Skow RJ, Meah VL, Riske L, Sobierajski F, James M, Kathol AJ, Nuspl M, Marchand AA, Nagpal TS, Slater LG, Weeks A, Adamo KB, Davies GA, Barakat R, Mottola MF. Prenatal exercise for the prevention of gestational diabetes mellitus and hypertensive disorders of pregnancy: a systematic review and meta-analysis. Br J Sports Med. 2018 Nov;52(21):1367-1375. doi: 10.1136/bjsports-2018-099355. PMID 30337463
- [Background] Genest DS, Falcao S, Gutkowska J, Lavoie JL. Impact of exercise training on preeclampsia: potential preventive mechanisms. Hypertension. 2012 Nov;60(5):1104-9. doi: 10.1161/HYPERTENSIONAHA.112.194050. Epub 2012 Oct 8. PMID 23045469
- [Background] Ferraro ZM, Gaudet L, Adamo KB. The potential impact of physical activity during pregnancy on maternal and neonatal outcomes. Obstet Gynecol Surv. 2012 Feb;67(2):99-110. doi: 10.1097/OGX.0b013e318242030e. PMID 22325300